CLINICAL TRIAL: NCT05840016
Title: A Randomized, Controlled, Multi-center Phase III Clinical Study of AK112 Combined With Chemotherapy Versus PD-1 Inhibitor Combined With Chemotherapy as First-line Treatment for Locally Advanced or Metastatic Squamous Non-small Cell Lung Cancer
Brief Title: AK112 in Combination With Chemotherapy in Advanced Squamous Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK112-306
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Advanced Squamous Non Small Cell Lung Cancer
MeSH Terms: interventions — Carboplatin; tislelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: AK112 in Combination With Paclitaxel Plus Carboplatin (Experimental): AK112 will be administered at a selected dose intravenously (IV) every three weeks (Q3W). Carboplatin will be administered at AUC5, Q3W, intravenously (IV) for 4 cycles. Paclitaxel will be administered at 175 mg/m2, Q3W, intravenously (IV) for 4 cycles.
  Interventions: Drug: AK112, Carboplatin, Paxlitaxel
- Active Comparator: Tislelizumab in Combination With Paclitaxel Plus Carboplatin (Active Comparator): Tislelizumab will be administered at a dose of 200 mg intravenously (IV) every three weeks (Q3W). Carboplatin will be administered at AUC5, Q3W, intravenously (IV) for 4 cycles. Paclitaxel will be administered at 175 mg/m2, Q3W, intravenously (IV) for 4 cycles.
  Interventions: Drug: Tislelizumab, Carboplatin, Paxlitaxel

INTERVENTIONS:
Drug: AK112, Carboplatin, Paxlitaxel — IV infusion,Specified dose on specified days
  Arms: Experimental: AK112 in Combination With Paclitaxel Plus Carboplatin
Drug: Tislelizumab, Carboplatin, Paxlitaxel — IV infusion,Specified dose on specified days
  Arms: Active Comparator: Tislelizumab in Combination With Paclitaxel Plus Carboplatin

SUMMARY:
This trial is a Phase III study. All patients are stage IIIB/C (unsuitable for radical therapy) or stage IV squamous non-small cell lung cancer(NSCLC), Eastern Cooperative Oncology Group (ECOG) performance status 0-1. The purpose of this study is to evaluate the efficacy and safety of AK112 combined with chemotherapy versus Tislelizumab combined with chemotherapy in patients with advanced squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).
* ≥18 years old and ≤75 years old (at the time consent is obtained).
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has a life expectancy of at least 3 months.
* Has a histologically confirmed diagnosis of squamous NSCLC.
* Has Stage IIIB/C or IV NSCLC (American Joint Committee on Cancer [AJCC]).
* Has no prior systemic anti-tumor therapy for locally advanced or metastatic NSCLC.
* Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Has adequate organ function.

Exclusion Criteria:

* Histological diagnosis of non-squamous NSCLC.
* Has EGFR-sensitive mutations or ALK gene translocations.
* Known ROS1 rearrangement, MET exon 14 skipping mutation, or RET gene fusion positivite.
* Is currently participating in a study of an investigational agent or using an investigational device.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy within 2 years prior to the first dose of study treatment.
* Has undergone major surgery within 30 days of Study Day 1.
* Has known active central nervous system (CNS) metastases.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has an active infection requiring systemic therapy.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* History of myocardial infarction, unstable angina, congestive heart failure within 12 months prior to day 1 of study treatment.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Has received a live virus vaccine within 30 days of the planned first dose of study therapy.
* Has any concurrent medical condition that, in the opinion of the Investigator, would complicate or compromise compliance with the study or the well-being of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS assessed by IRRC per RECIST v1.1 | Up to approximately 2 years
  Progression-free survival (PFS) is defined as the time from the date of randomization till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the blinded IRRC or death due to any cause (whichever occurs first).

SECONDARY OUTCOMES:
OS | Up to approximately 2 years
  Overall Survival (OS) is defined as the time from the start of treatment with AK112 until death due to any cause.
ORR assessed by IRRC per RECIST v1.1 | Up to approximately 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on RECIST v1.1.
DoR assessed by IRRC per RECIST v1.1 | Up to approximately 2 years
  Duration of response (DoR) assessed according to RECIST v1.1
DCR assessed by IRRC per RECIST v1.1 | Up to approximately 2 years
  Disease control rate (DCR) assessed according to RECIST v1.1.
TTR assessed by IRRC per RECIST v1.1 | Up to approximately 2 years
  Time to response (TTR) is defined as the time to response base on RECIST v1.1.
PFS assessed by investigator per RECIST v1.1 | Up to approximately 2 years
  Progression-free survival (PFS) is defined as the time from the date of randomization till the first documentation of disease progression assessed by the investigator or death due to any cause (whichever occurs first).
ORR assessed by the investigator per RECIST v1.1 | Up to approximately 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on RECIST v1.1.
DoR assessed by the investigator per RECIST v1.1 | Up to approximately 2 years
  Duration of response (DoR) assessed according to RECIST v1.1.
DCR assessed by the investigator per RECIST v1.1 | Up to approximately 2 years
  Disease control rate (DCR) assessed according to RECIST v1.1.
TTR assessed by the investigator per RECIST v1.1 | Up to approximately 2 years
  Time to response (TTR) is defined as the time to response base on RECIST v1.1.
AE | Up to approximately 2 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
ADA | Up to approximately 2 years
  Number of subjects with detectable anti-drug antibodies (ADA).
Cmax and Cmin | Up to approximately 2 years
  AK112 serum drug concentrations in subjects at different time points after AK112 administration
PD-L1 expression | Up to approximately 2 years
  The correlationship between PD-L1 expression and efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China